CLINICAL TRIAL: NCT05964452
Title: The Efficacy of Cook County Health's Methimazole Dosing Algorithm in the Setting of Ne Onset Graves' Hyperthyroidism
Brief Title: Efficacy of Methimazole Dosing Algorithm
Status: Terminated | Type: Observational
Why Stopped: Unable to reach recruiting goals
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Dan Mihailescu, MD Endocrinology Cluster Director, Cook County Health
Other Study IDs: 22-010
Record Dates: First submitted 2023-07-17; First posted 2023-07-28 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: Graves Disease
MeSH Terms: conditions — Graves Disease | interventions — Methimazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Methimazole Tablets — Testing dosing algorithm for efficacy.
  Other Names: Tapazole

SUMMARY:
To prospectively study the efficacy and safety of the Cook County Health (CCH) methimazole (MMI) dosing algorithm in the setting of new onset Graves' disease.

DETAILED DESCRIPTION:
To conduct a prospective observational study in 60 patients with newly diagnosed Graves' disease who are either methimazole naive or who have been initiated on MMI within previous 4-6 weeks per CCH algorithm and assess for efficacy and safety of MMI dosing administered. Study group size is based on 90% power and projected efficacy of 70% patients reaching target.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adults (>18 years of age) with new diagnosis of Graves' Disease (elevated free T4, Free T3, low or suppressed TSH, positive TSI and or thyroid eye disease) and
* either drug naïve or who have been initiated on MMI within previous 4-6 weeks per CCH algorithm.

Exclusion Criteria:

* Pregnant patients
* hyperthyroidism due to other causes, example - Toxic Multinodular Goiter, Iodine induced thyrotoxicosis, etc.
* Graves patients who present with atrial fibrillation, CHF or other end organ damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with new onset Graves' disease.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Achievement of euthyroid state | 17 weeks
  The proportion of patients achieving euthyroid state during the study period

SECONDARY OUTCOMES:
Factors influencing achievement of euthyroid state | 17 weeks
  Identifying variables that correlate with achievement of euthyroid state

CONTACTS AND LOCATIONS:
Overall Officials: Dan Mihailescu, MD, Principal Investigator — Cook County Health
Locations (1):
- Cook County Health, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Study not completed